CLINICAL TRIAL: NCT06465628
Title: Effect of Self-administered Acupressure for Improving Xerostomia in Head and Neck Cancer Patients: a Randomized Controlled Trial
Brief Title: Acupressure on Xerostomia in Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-233
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Cancer; Xerostomia
Keywords: Self-administered acupressure; Xerostomia; Head and neck cancer; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Health Education, Dental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-administered acupressure (Experimental): Participants will attend a 90-min self-administered acupressure training session by a registered Traditional Chinese Medicine practitioner. A follow-up session will be arranged in the second week to reinforce learning and to make sure all participants can locate the proposed acupoints correctly. The follow up session will be conducted face to face (prioritized mode), or by phone/video call based on patients' preference. The acupoints are chosen for inclusion in the protocol based on literature review [25, 29, 34, 35, 39] and expert experience of the PI [40-43]. The location of acupoints (nine in total) include face and neck (Ren 23, Ren 24, ST5, ST6, ST7, TE17), upper limbs (LI2, LI4), and lower limbs (KI6). All acupoints should be massaged bilaterally except Ren 23 and Ren 24. After the training, participants are encouraged to self-administered acupressure on the acupoints twice daily for 12 weeks, each point lasting for 1 minute.
  Interventions: Behavioral: Self-administered acupressure
- Oral health education (Active Comparator): Participants will attend a 90-min oral care education session in the first week by a trained research staff (the same frequency and duration as the intervention group). The content includes the causes of xerostomia, consequences, current preventative measures, dietary advice and oral hygiene advice.
  Participants in the control group will receive a booklet documenting the content of the oral care education sessions. Throughout the 12-week period, participants will receive reminders of oral care for xerostomia twice weekly
  Interventions: Other: Oral health education

INTERVENTIONS:
Behavioral: Self-administered acupressure — The participants should perform self-administered acupressure 12 weeks after training
  Arms: Self-administered acupressure
Other: Oral health education — The participants should perform general oral care by themselves after the oral health education relating to xerostomia
  Arms: Oral health education

SUMMARY:
This is a randomized controlled trial aimed to1) examine the effect of a self-administered acupressure intervention on head and neck cancer patients with xerostomia (primary outcome) relative to oral health education control; 2) examine the effect of self-administered acupressure on secondary outcomes, including quality of life and severity of symptoms of head and neck cancer patients; 3) evaluate patients' expectancy of acupressure; 4) explore the acceptability of self-administered acupressure for head and neck cancer patients with xerostomia.

Hypothesis: self-administered acupressure has better effect on xerostomia for head and neck cancer patients comparing to oral health education. Acupressure will also benefit head and neck cancer patients on quality of life and severity of symptoms. Head and neck cancer patients may have good acceptability of self-administered acupressure.

DETAILED DESCRIPTION:
Xerostomia is defined as "the subjective sensation of dryness of the mouth". It is common in patients with acute/chronic medical conditions, especially in patients with cancer. Results from observational studies reported 40% to 75% prevalence of xerostomia among cancer patients. Head and neck cancer patients, as the seventh most common type of cancer, reported an even higher prevalence (80%) of xerostomia after treatment compared with other cancer types. Despite the high prevalence of xerostomia, it is often underrecognized by patients and healthcare providers.

Xerostomia in head and neck cancer patients is largely induced by radiation in the head and neck region, which can damage salivary glands, and thereby change the volume, consistency, and pH of their saliva. Besides, xerostomia may be caused or exacerbated by the concomitant or sequential use of chemotherapy agents and other drugs (e.g., opioid). Consistent lacking saliva in cancer patients can lead to increased risk of oral fungal infection, caries, swallowing problems, sleep problems, depression, fatigue and altered taste, which may even result in poor nutritional status. Furthermore, xerostomia may become a chronic and even irreversible side effect.

Current therapies for xerostomia in cancer patients include both pharmacological and non-pharmacological treatments. Pharmacotherapy has been considered as a general treatment for stimulating saliva secretion in alleviating xerostomia for head and neck cancer patients. However, the evidence of pharmacological interventions (e.g., pilocarpine, bethanechol, amifostin, cevimeline and palifermin) on xerostomia is insufficient, and the use of pharmacotherapy may cause some common adverse effects, including nausea, sweating, nervousness, and urinary frequency. Non-pharmacological treatments such as saliva stimulants (e.g. citric and malic acids, chewing gum, toothpaste and lozenges) and saliva substitute (e.g. liquids, gels and sprays) have also been suggested to treat xerostomia, but neither with sufficient evidence of significant effect, and may also lead to adverse effects (e.g., nausea, unpleasant taste, diarrhea, and tooth mineralization). Some patients may find regular sips of water useful, but only for temporary benefit, because saliva is a complex substance with irreplaceable functions (antibacterial and immunologic protection). Therefore, an evidence-based effective strategy with few adverse events is warranted for head and neck cancer patients with xerostomia.

Both acupressure and acupuncture aim to improve health and cure illnesses by improving energy flow through stimulating meridian points. Acupressure is a non-invasive technique of activating acupoints using hands, fingers, or thumbs along the meridians, while acupuncture involves the use of needles. Stimulation on acupoints may increase the flow of blood and qi along the related meridians, as well as stimulate the local blood flow around the salivary glands, thereby increasing salivary secretion. Also, acupressure/acupuncture may stimulate the parasympathetic nervous system, hence indirectly stimulate salivary glands secretion. Besides, microcirculation may be promoted through the release of sensory neuropeptides, so as to increase the tissue oxygenation and metabolism. Some studies had demonstrated positive effect of acupuncture on xerostomia for head and neck cancer patients, while none examined acupressure. Based on the same meridian theory, both acupuncture and acupressure were widely applied to the symptom management (e.g. fatigue, nausea, pain) for cancer patients, effectively with good adherence. Compared to acupuncture, acupressure can be administered by patients themselves after training. The purpose of this study is to examine the effect of self-administered acupressure on xerostomia for head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* able to give informed consent;
* diagnosed with head and neck cancer (cancers in the head and neck region, e.g. oral cancer, nasopharyngeal cancer, oropharyngeal cancer, hypopharyngeal cancer, laryngeal cancer, sinus cancer, salivary gland cancer);
* completed radiation therapy or chemoradiotherapy for at least 2 weeks;
* complains of xerostomia after the treatment;
* able to communicate in Cantonese or Mandarin.

Exclusion Criteria:

* history of xerostomia prior to head and neck cancer treatment (e.g., Sjögren Syndrome);
* practiced acupressure or received acupuncture in the last 3 months;
* having contraindications to acupressure, e.g. blood system disease (e.g., leukemia); pregnancy; lactating; upper or lower extremity deformities; infection or injuries at the acupoints.

Those who are taking medications/alternative substances to treat xerostomia on a fixed dosage regimen in the past one month will not be excluded.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Xerostomia Questionnaire | Baseline, 4 weeks, 12 weeks, and 24 weeks
  Self-reported severity of xerostomia will be measured using the Xerostomia Questionnaire at baseline, 4 weeks, 12 weeks and 24 weeks. It consists of 8 items on an 11-point scale (0-80), which has been validated in several cohorts, and is regarded as the criterion standard for measuring xerostomia, which has been used for patients with head and neck cancer. Higher score refers to higher level in xerostomia. After adding item scores, the sum is transformed linearly to produce a final summary score between 0 and 100. Higher scores represent higher level of xerostomia. It suggested that an XQ score ≤30 refers to mild to no symptoms of xerostomia.

SECONDARY OUTCOMES:
Saliva flow | baseline, 12 weeks and 24 weeks
  Objectively measured severity of xerostomia will be measured using modified Schirmer strips between 9 am to 12 pm. The modified Schirmer test is an objective, well-tolerated test for measuring mouth dryness for head and neck cancer patients. Before performing the test, all the participants should refrain from eating and drinking for at least 15 min. The participants will be asked to swallow once before the measurement. Unstimulated saliva will be measured by inserting a test strip to the floor of the mouth for three minutes (remove the strip for two to three second and to read the test strip at 1-minute, 2-minute and 3-minute respectively, with one-minute interval between each reading). Then, patients will have fresh lemon juice applied with cotton-tipped applicators to the lateral tongue bilaterally five times(apply at 0, 30s, 60s, 90s and 120s respectively). The stimulated saliva will be collected in the same manner as for unstimulated saliva
Quality of life for head and neck cancer patients | baseline, 12 weeks and 24 weeks
  European Organisation for Research and Treatment of Cancer Quality of Life-Head and Neck cancer (EORTC QLQ-HN35) will be used to estimate the quality of life for head and neck cancer patients. The standardized sum scores range from 0 to 100, with a higher score indicating a greater degree of symptoms (worse QOL)
Symptom severity | baseline, 12 weeks and 24 weeks
  MD Anderson Symptom Inventory-Head and Neck (MDASI-HN) will be used to measure the severity of different cancer symptoms and the interference of symptoms with patients' daily activities at baseline, 12 weeks and 24 weeks. MDASI-HN consists of 28 items, and the range of scores is 0-280, with a higher degree indicating a greater degree of symptoms. The scale has been validated in studies evaluating symptom severity and daily activities for head and neck cancer patients.
Sociodemographic characteristics | Baseline
  The sociodemographic characteristics will be collected at baseline, such as age, gender, education levels, employment, marital status (single/married/cohabitating/divorced), income levels, smoking/drinking status, comorbidities, cancer types, cancer stage, cancer treatment, and time since finishing the cancer treatment.
Acceptability | 12 week
  Acceptability of the intervention will be measured in terms of training and self-practice adherence. Training adherence is defined as the percentage of patients who completed the two intervention sessions. Self-practice adherence is defined as the proportion of participants completing more than 70% of prescribed self-practice. Overall adherence is defined as the proportion of participants completing the two intervention sessions and more than 70% of prescribed self-practice
Acupressure Expectancy Scale | Baseline
  The Acupressure Expectancy Scale consists of 4 items using a five-point scale, with higher score indicating higher expectations (score range, 0-16)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Cheung, PhD, Principal Investigator — School of Nursing, the University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
We are not to share IPD. All IPD for patients will be collected and analyzed confidentially, they can only be identified with their unique ID in this study. Only members in this research team have access to the personal and study data during the validity period. The PI will be responsible for safekeeping of the study data.

REFERENCES:
- [Background] Davies AN. A comparison of artificial saliva and chewing gum in the management of xerostomia in patients with advanced cancer. Palliat Med. 2000 May;14(3):197-203. doi: 10.1191/026921600672294077. PMID 10858827
- [Background] Eisbruch A, Kim HM, Terrell JE, Marsh LH, Dawson LA, Ship JA. Xerostomia and its predictors following parotid-sparing irradiation of head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Jul 1;50(3):695-704. doi: 10.1016/s0360-3016(01)01512-7. PMID 11395238
- [Background] Jensen SB, Pedersen AM, Vissink A, Andersen E, Brown CG, Davies AN, Dutilh J, Fulton JS, Jankovic L, Lopes NN, Mello AL, Muniz LV, Murdoch-Kinch CA, Nair RG, Napenas JJ, Nogueira-Rodrigues A, Saunders D, Stirling B, von Bultzingslowen I, Weikel DS, Elting LS, Spijkervet FK, Brennan MT; Salivary Gland Hypofunction/Xerostomia Section, Oral Care Study Group, Multinational Association of Supportive Care in Cancer (MASCC)/International Society of Oral Oncology (ISOO). A systematic review of salivary gland hypofunction and xerostomia induced by cancer therapies: prevalence, severity and impact on quality of life. Support Care Cancer. 2010 Aug;18(8):1039-60. doi: 10.1007/s00520-010-0827-8. Epub 2010 Mar 17. PMID 20237805
- [Background] Mercadante S, Calderone L, Villari P, Serretta R, Sapio M, Casuccio A, Fulfaro F. The use of pilocarpine in opioid-induced xerostomia. Palliat Med. 2000 Nov;14(6):529-31. doi: 10.1191/026921600701536273. No abstract available. PMID 11219883
- [Background] Garcia-Chias B, Figuero E, Castelo-Fernandez B, Cebrian-Carretero JL, Cerero-Lapiedra R. Prevalence of oral side effects of chemotherapy and its relationship with periodontal risk: a cross sectional study. Support Care Cancer. 2019 Sep;27(9):3479-3490. doi: 10.1007/s00520-019-4650-6. Epub 2019 Jan 24. PMID 30675665
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Nathan CO, Asarkar AA, Entezami P, Corry J, Strojan P, Poorten VV, Makitie A, Eisbruch A, Robbins KT, Smee R, St John M, Chiesa-Estomba C, Winter SC, Beitler JJ, Ferlito A. Current management of xerostomia in head and neck cancer patients. Am J Otolaryngol. 2023 Jul-Aug;44(4):103867. doi: 10.1016/j.amjoto.2023.103867. Epub 2023 Mar 28. PMID 36996514
- [Background] Dirix P, Nuyts S, Vander Poorten V, Delaere P, Van den Bogaert W. The influence of xerostomia after radiotherapy on quality of life: results of a questionnaire in head and neck cancer. Support Care Cancer. 2008 Feb;16(2):171-9. doi: 10.1007/s00520-007-0300-5. Epub 2007 Jul 6. PMID 17618467
- [Background] Bhide SA, Miah AB, Harrington KJ, Newbold KL, Nutting CM. Radiation-induced xerostomia: pathophysiology, prevention and treatment. Clin Oncol (R Coll Radiol). 2009 Dec;21(10):737-44. doi: 10.1016/j.clon.2009.09.002. Epub 2009 Oct 14. PMID 19833490
- [Background] Chambers MS, Garden AS, Kies MS, Martin JW. Radiation-induced xerostomia in patients with head and neck cancer: pathogenesis, impact on quality of life, and management. Head Neck. 2004 Sep;26(9):796-807. doi: 10.1002/hed.20045. PMID 15350026
- [Background] Walsh M, Fagan N, Davies A. Xerostomia in patients with advanced cancer: a scoping review of clinical features and complications. BMC Palliat Care. 2023 Nov 11;22(1):178. doi: 10.1186/s12904-023-01276-4. PMID 37950188
- [Background] Porter SR, Scully C, Hegarty AM. An update of the etiology and management of xerostomia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Jan;97(1):28-46. doi: 10.1016/j.tripleo.2003.07.010. PMID 14716254
- [Background] Bustillos H, Indorf A, Alwan L, Thompson J, Jung L. Xerostomia: an immunotherapy-related adverse effect in cancer patients. Support Care Cancer. 2022 Feb;30(2):1681-1687. doi: 10.1007/s00520-021-06535-9. Epub 2021 Sep 25. PMID 34562169
- [Background] Warner BM, Baer AN, Lipson EJ, Allen C, Hinrichs C, Rajan A, Pelayo E, Beach M, Gulley JL, Madan RA, Feliciano J, Grisius M, Long L, Powers A, Kleiner DE, Cappelli L, Alevizos I. Sicca Syndrome Associated with Immune Checkpoint Inhibitor Therapy. Oncologist. 2019 Sep;24(9):1259-1269. doi: 10.1634/theoncologist.2018-0823. Epub 2019 Apr 17. PMID 30996010
- [Background] Moral Nakamura D, da Graca Pinto H, Baena Elchin C, Thomazotti Berard L, Abreu Alves F, Azeredo Alves Antunes L, Pena Coto N. Efficacy of bethanechol chloride in the treatment of radiation-induced xerostomia in patients with head and neck cancer: A systematic review and meta-analysis. Radiother Oncol. 2023 Sep;186:109715. doi: 10.1016/j.radonc.2023.109715. Epub 2023 May 18. PMID 37207874
- [Background] Cheng CQ, Xu H, Liu L, Wang RN, Liu YT, Li J, Zhou XK. Efficacy and safety of pilocarpine for radiation-induced xerostomia in patients with head and neck cancer: A systematic review and meta-analysis. J Am Dent Assoc. 2016 Apr;147(4):236-43. doi: 10.1016/j.adaj.2015.09.014. Epub 2015 Nov 10. PMID 26563850
- [Background] Yang WF, Liao GQ, Hakim SG, Ouyang DQ, Ringash J, Su YX. Is Pilocarpine Effective in Preventing Radiation-Induced Xerostomia? A Systematic Review and Meta-analysis. Int J Radiat Oncol Biol Phys. 2016 Mar 1;94(3):503-11. doi: 10.1016/j.ijrobp.2015.11.012. Epub 2015 Nov 10. PMID 26867879
- [Background] Riley P, Glenny AM, Hua F, Worthington HV. Pharmacological interventions for preventing dry mouth and salivary gland dysfunction following radiotherapy. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD012744. doi: 10.1002/14651858.CD012744. PMID 28759701
- [Background] Mercadante S, Aielli F, Adile C, Ferrera P, Valle A, Fusco F, Caruselli A, Cartoni C, Massimo P, Masedu F, Valenti M, Porzio G. Prevalence of oral mucositis, dry mouth, and dysphagia in advanced cancer patients. Support Care Cancer. 2015 Nov;23(11):3249-55. doi: 10.1007/s00520-015-2720-y. Epub 2015 Apr 3. PMID 25832897
- [Background] Kahn ST, Johnstone PA. Management of xerostomia related to radiotherapy for head and neck cancer. Oncology (Williston Park). 2005 Dec;19(14):1827-32; discussion 1832-4, 1837-9. PMID 16506635
- [Background] Hahnel S, Behr M, Handel G, Burgers R. Saliva substitutes for the treatment of radiation-induced xerostomia--a review. Support Care Cancer. 2009 Nov;17(11):1331-43. doi: 10.1007/s00520-009-0671-x. Epub 2009 Jun 4. PMID 19495809
- [Background] Bots CP, Brand HS, Veerman EC, Valentijn-Benz M, Van Amerongen BM, Nieuw Amerongen AV, Valentijn RM, Vos PF, Bijlsma JA, Bezemer PD, ter Wee PM. The management of xerostomia in patients on haemodialysis: comparison of artificial saliva and chewing gum. Palliat Med. 2005 Apr;19(3):202-7. doi: 10.1191/0269216305pm1009oa. PMID 15920934
- [Background] Assery MKA. Efficacy of Artificial Salivary Substitutes in Treatment of Xerostomia: A Systematic Review. J Pharm Bioallied Sci. 2019 Feb;11(Suppl 1):S1-S12. doi: 10.4103/jpbs.JPBS_220_18. PMID 30923424
- [Background] Liu G, Qiu X, Tan X, Miao R, Tian W, Jing W. Efficacy of a 1% malic acid spray for xerostomia treatment: A systematic review and meta-analysis. Oral Dis. 2023 Apr;29(3):862-872. doi: 10.1111/odi.14116. Epub 2022 Jan 17. PMID 34954846
- [Background] Assy Z, Brand HS. A systematic review of the effects of acupuncture on xerostomia and hyposalivation. BMC Complement Altern Med. 2018 Feb 13;18(1):57. doi: 10.1186/s12906-018-2124-x. PMID 29439690
- [Background] Momm F, Volegova-Neher NJ, Schulte-Monting J, Guttenberger R. Different saliva substitutes for treatment of xerostomia following radiotherapy. A prospective crossover study. Strahlenther Onkol. 2005 Apr;181(4):231-6. doi: 10.1007/s00066-005-1333-7. PMID 15827692
- [Background] Blom M, Dawidson I, Fernberg JO, Johnson G, Angmar-Mansson B. Acupuncture treatment of patients with radiation-induced xerostomia. Eur J Cancer B Oral Oncol. 1996 May;32B(3):182-90. doi: 10.1016/0964-1955(95)00085-2. PMID 8762876
- [Background] Naik PN, Kiran RA, Yalamanchal S, Kumar VA, Goli S, Vashist N. Acupuncture: An Alternative Therapy in Dentistry and Its Possible Applications. Med Acupunct. 2014 Dec 1;26(6):308-314. doi: 10.1089/acu.2014.1028. PMID 25538815
- [Background] Meng Z, Kay Garcia M, Hu C, Chiang J, Chambers M, Rosenthal DI, Peng H, Wu C, Zhao Q, Zhao G, Liu L, Spelman A, Lynn Palmer J, Wei Q, Cohen L. Sham-controlled, randomised, feasibility trial of acupuncture for prevention of radiation-induced xerostomia among patients with nasopharyngeal carcinoma. Eur J Cancer. 2012 Jul;48(11):1692-9. doi: 10.1016/j.ejca.2011.12.030. Epub 2012 Jan 28. PMID 22285177
- [Background] Meng Z, Garcia MK, Hu C, Chiang J, Chambers M, Rosenthal DI, Peng H, Zhang Y, Zhao Q, Zhao G, Liu L, Spelman A, Palmer JL, Wei Q, Cohen L. Randomized controlled trial of acupuncture for prevention of radiation-induced xerostomia among patients with nasopharyngeal carcinoma. Cancer. 2012 Jul 1;118(13):3337-44. doi: 10.1002/cncr.26550. Epub 2011 Nov 9. PMID 22072272
- [Background] Simcock R, Fallowfield L, Monson K, Solis-Trapala I, Parlour L, Langridge C, Jenkins V; ARIX Steering Committee. ARIX: a randomised trial of acupuncture v oral care sessions in patients with chronic xerostomia following treatment of head and neck cancer. Ann Oncol. 2013 Mar;24(3):776-83. doi: 10.1093/annonc/mds515. Epub 2012 Oct 25. PMID 23104718
- [Background] Pfister DG, Cassileth BR, Deng GE, Yeung KS, Lee JS, Garrity D, Cronin A, Lee N, Kraus D, Shaha AR, Shah J, Vickers AJ. Acupuncture for pain and dysfunction after neck dissection: results of a randomized controlled trial. J Clin Oncol. 2010 May 20;28(15):2565-70. doi: 10.1200/JCO.2009.26.9860. Epub 2010 Apr 20. PMID 20406930
- [Background] Garcia MK, Meng Z, Rosenthal DI, Shen Y, Chambers M, Yang P, Wei Q, Hu C, Wu C, Bei W, Prinsloo S, Chiang J, Lopez G, Cohen L. Effect of True and Sham Acupuncture on Radiation-Induced Xerostomia Among Patients With Head and Neck Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1916910. doi: 10.1001/jamanetworkopen.2019.16910. PMID 31808921
- [Background] Ni X, Tian T, Chen D, Liu L, Li X, Li F, Liang F, Zhao L. Acupuncture for Radiation-Induced Xerostomia in Cancer Patients: A Systematic Review and Meta-Analysis. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420980825. doi: 10.1177/1534735420980825. PMID 33307864
- [Background] de Sousa TR, Mattos S, Marcon G, Furtado T, Duarte da Silva M. Acupuncture techniques and acupoints used in individuals under chemotherapy or radiotherapy treatment of cancer: A systematic review. J Clin Nurs. 2023 Oct;32(19-20):6917-6933. doi: 10.1111/jocn.16812. Epub 2023 Jun 29. PMID 37382085
- [Background] He Y, Guo X, May BH, Zhang AL, Liu Y, Lu C, Mao JJ, Xue CC, Zhang H. Clinical Evidence for Association of Acupuncture and Acupressure With Improved Cancer Pain: A Systematic Review and Meta-Analysis. JAMA Oncol. 2020 Feb 1;6(2):271-278. doi: 10.1001/jamaoncol.2019.5233. PMID 31855257
- [Background] Lau CHY, Wu X, Chung VCH, Liu X, Hui EP, Cramer H, Lauche R, Wong SYS, Lau AYL, Sit RWS, Ziea ETC, Ng BFL, Wu JCY. Acupuncture and Related Therapies for Symptom Management in Palliative Cancer Care: Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 Mar;95(9):e2901. doi: 10.1097/MD.0000000000002901. PMID 26945382
- [Background] Cheng HL, Yeung WF, Wong HF, Lo HT, Molassiotis A. Self-Acupressure for Symptom Management in Cancer Patients: A Systematic Review. J Pain Symptom Manage. 2023 Jul;66(1):e109-e128. doi: 10.1016/j.jpainsymman.2023.03.002. Epub 2023 Mar 9. PMID 36898639
- [Background] Braga FP, Lemos Junior CA, Alves FA, Migliari DA. Acupuncture for the prevention of radiation-induced xerostomia in patients with head and neck cancer. Braz Oral Res. 2011 Mar-Apr;25(2):180-5. doi: 10.1590/s1806-83242011000200014. PMID 21537645
- [Background] Cheung DST, Tiwari A, Yeung WF, Yu DSF, So MKP, Chau PH, Wang XM, Lum TYS, Yuk Fung HYK, Ng BYM, Zhang ZJ, Lao L. Self-Administered Acupressure for Caregivers of Older Family Members: A Randomized Controlled Trial. J Am Geriatr Soc. 2020 Jun;68(6):1193-1201. doi: 10.1111/jgs.16357. Epub 2020 Feb 25. PMID 32096884
- [Background] Cheung DST, Yeung WF, Suen LK, Chong TC, Ho YS, Yu BY, Chan LY, Chen HY, Lao LX. Self-administered acupressure for knee osteoarthritis in middle-aged and older adults: a pilot randomized controlled trial. Acupunct Med. 2020 Apr;38(2):75-85. doi: 10.1177/0964528419883269. Epub 2019 Nov 13. PMID 31718229
- [Background] Cheung DST, Yeung WF, Chau PH, Lam TC, Yang M, Lai K, Ip CY, Lao L, Lin CC. Patient-centred, self-administered acupressure for Chinese advanced cancer patients experiencing fatigue and co-occurring symptoms: A pilot randomised controlled trial. Eur J Cancer Care (Engl). 2022 Sep;31(5):e13314. doi: 10.1111/ecc.13314. Epub 2020 Sep 7. PMID 32896014
- [Background] Cheung DST, Xu X, Smith R, Takemura N, Yeung WF, Chan WL, Lao L, Lin CC. Invasive or noninvasive? A systematic review and network meta-analysis of acupuncture and acupressure to treat sleep disturbance in cancer patients. Worldviews Evid Based Nurs. 2023 Jun;20(3):202-211. doi: 10.1111/wvn.12617. Epub 2022 Dec 21. PMID 36541042
- [Background] Huang SH, de Almeida JR, Watson E, Glogauer M, Xu W, Keshavarzi S, O'Sullivan B, Ringash J, Hope A, Bayley A, Bratman SV, Cho J, Giuliani M, Kim J, Waldron J, Spreafico A, Goldstein DP, Chepeha DB, Li T, Hosni A. Short-term and long-term unstimulated saliva flow following unilateral vs bilateral radiotherapy for oropharyngeal carcinoma. Head Neck. 2021 Feb;43(2):456-466. doi: 10.1002/hed.26496. Epub 2020 Oct 15. PMID 33058305
- [Background] Deboni AL, Giordani AJ, Lopes NN, Dias RS, Segreto RA, Jensen SB, Segreto HR. Long-term oral effects in patients treated with radiochemotherapy for head and neck cancer. Support Care Cancer. 2012 Nov;20(11):2903-11. doi: 10.1007/s00520-012-1418-7. Epub 2012 Mar 13. PMID 22410861
- [Background] Lal P, Bajpai R, Khurana R, Das KJ, Kumar P, Tiwari A, Gupta N, Kumar S. Changes in salivary flow rates in head and neck cancer after chemoradiotherapy. J Cancer Res Ther. 2010 Oct-Dec;6(4):458-62. doi: 10.4103/0973-1482.77105. PMID 21358080
- [Background] EORTC. European Organisation for Research and Treatment of Cancer Quality of life-head and neck cancer 1994 [cited 2023 Dec]; Available from: https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-HN35-English.pdf.
- [Background] Aarstad HJ, Osthus AA, Aarstad HH, Lybak S, Aarstad AKH. EORTC Quality of Life Questionnaire Head and Neck (H&N)-35 scores from H&N squamous cell carcinoma patients obtained at diagnosis and at 6, 9 and 12 months following diagnosis predict 10-year overall survival. Eur Arch Otorhinolaryngol. 2019 Dec;276(12):3495-3505. doi: 10.1007/s00405-019-05630-2. Epub 2019 Sep 16. PMID 31529149
- [Background] Bjordal K, Ahlner-Elmqvist M, Tollesson E, Jensen AB, Razavi D, Maher EJ, Kaasa S. Development of a European Organization for Research and Treatment of Cancer (EORTC) questionnaire module to be used in quality of life assessments in head and neck cancer patients. EORTC Quality of Life Study Group. Acta Oncol. 1994;33(8):879-85. doi: 10.3109/02841869409098450. PMID 7818919
- [Background] Rosenthal DI, Mendoza TR, Chambers MS, Asper JA, Gning I, Kies MS, Weber RS, Lewin JS, Garden AS, Ang KK, S Wang X, Cleeland CS. Measuring head and neck cancer symptom burden: the development and validation of the M. D. Anderson symptom inventory, head and neck module. Head Neck. 2007 Oct;29(10):923-31. doi: 10.1002/hed.20602. PMID 17358040
- [Background] Mao JJ, Xie SX, Bowman MA. Uncovering the expectancy effect: the validation of the acupuncture expectancy scale. Altern Ther Health Med. 2010 Nov-Dec;16(6):22-7. PMID 21280459